CLINICAL TRIAL: NCT00732056
Title: A Phase I/II Study of GRN163L in Combination With Paclitaxel and Bevacizumab in Patients With Locally Recurrent or Metastatic Breast Cancer
Brief Title: A Study of GRN163L With Paclitaxel and Bevacizumab to Treat Patients With Locally Recurrent Or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRN163L CP14A010
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer; Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — GRN163L peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 3+3 cohort dose escalation
  Interventions: Drug: GRN163L

INTERVENTIONS:
Drug: GRN163L — 25% dose escalation infused over 2 hours weekly

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of GRN163L in combination with paclitaxel and bevacizumab in patients with locally recurrent or metastatic breast cancer (MBC)

DETAILED DESCRIPTION:
GRN163L is a telomerase template antagonist with in vitro and in vivo activity in a variety of tumor model systems. Telomerase is an enzyme that is active primarily in tumor cells and is crucial for the indefinite growth of tumor cells. Inhibition of telomerase may result in antineoplastic effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with measurable locally recurrent or metastatic disease
* May have had one prior non-taxane chemotherapy regimen for metastatic disease
* If HER2 positive, must have had prior treatment with trastuzumab (Herceptin®)
* If previously treated with an anthracycline, anthracenedione, or trastuzumab must be tested by MUGA scan or echocardiogram and have LVEF ≥ 50%
* Must have recovered from most recent radiation treatment or surgical procedure
* ECOG performance status of 0 or 1
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Locally recurrent disease amenable to resection with curative intent
* Prior adjuvant or neoadjuvant taxane chemotherapy within 12 months prior to first study drug administration
* Investigational therapy within 4 weeks prior to first study drug administration
* Prior hormonal therapy within 2 weeks prior to first study drug administration
* Prior radiotherapy within 2 weeks prior to first study drug administration
* Cytotoxic chemotherapy within 2 weeks prior to first study drug administration
* Therapeutic anticoagulation or regular use of anti-platelet therapy within 2 weeks prior to first study drug administration NOTE: Low-dose anticoagulant therapy to maintain patency of a vascular access device is allowed.
* Prolongation of PT or INR, aPTT > ULN, or fibrinogen < LLN
* Active or chronically current bleeding (eg, active peptic ulcer)
* Clinically significant cardiovascular or cerebrovascular disease including

Any history of:

* Cerebrovascular disease including TIA, stroke or subarachnoid hemorrhage
* Ischemic bowel

Within the last 12 months:

* MI
* Unstable angina
* NYHA grade II or greater CHF
* Grade 2 or greater peripheral vascular disease

Active at study entry:

* Uncontrolled hypertension defined as SBP > 160 or DBP > 90
* Uncontrolled or clinically significant arrhythmia
* Clinically relevant active infection
* Nonhealing wound or fracture
* Serious co-morbid medical conditions, including cirrhosis and chronic obstructive or chronic restrictive pulmonary disease
* Active autoimmune disease requiring immunosuppressive therapy
* Known positive serology for HIV
* Prior malignancy (within the last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, or in situ prostate cancer, or other cancer for which the patient has been disease-free for at least 3 years
* Any other severe, acute, or chronic medical or psychiatric condition, laboratory abnormality, or difficult complying with protocol requirements that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety, MTD, efficacy | First 4 weeks

SECONDARY OUTCOMES:
PK and efficacy | Baseline to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (2):
- United States (2):
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

REFERENCES:
- See also: Related Info — http://www.geron.com